CLINICAL TRIAL: NCT00067522
Title: Family Planning Promotion to Prevent Unplanned Pregnancies in HIV Infected Zambian Couples
Brief Title: Preventing Unplanned Pregnancies in HIV Infected Zambian Couples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HD40125; 1R01HD040125-01A1 (NIH)
Record Dates: First submitted 2003-08-21; First posted 2003-08-25 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2005-09

CONDITIONS: Pregnancy; HIV Infections
Keywords: Family Planning; Sexually Transmitted Diseases; HIV; Africa; Zambia; AIDS; Contraception; HIV Prevention
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Behavioral: User-independent contraception program
Behavioral: Future Planning Perspectives program

SUMMARY:
Prevention of unplanned pregnancies among HIV infected couples decreases the rate of maternal-child virus transmission and the number of children orphaned when parents die of AIDS. This study will evaluate two programs for reducing the number of unplanned pregnancies among HIV infected couples in Zambia.

DETAILED DESCRIPTION:
Eighty percent of the world's HIV infections are in sub-Saharan Africa. In Lusaka, the capital of Zambia, 85% of pregnant women are married and 47% are in couples with at least one HIV infected partner (26% concordant positive, 21% discordant). It will be years before short-course antivirals are widely implemented, and many children who escape infection will be left orphaned. There are 360,000 AIDS orphans in Zambia, a country of 9 million people, and 35,000 HIV infected women deliver each year.

An essential component of any HIV prevention strategy must include the prevention of unplanned pregnancies among couples with HIV. Promotion of 'dual method' contraception (condoms for HIV/STD prevention plus a longer acting method for pregnancy prevention) is ideal, but unfortunately not widely promoted. Ultimately, the prevention of unplanned pregnancy in couples with HIV can reduce pediatric HIV, AIDS orphans, and the family consequences of parental illness and death.

This study will evaluate two interventions aimed at reducing the incidence of unplanned pregnancies in HIV infected couples. The first intervention will promote more effective contraception by placing user-independent methods (IUD and Norplant) first in the educational message hierarchy (currently, family planning education highlights oral contraceptives) and employing positive message framing. The second intervention will help couples plan for the consequences of their illness and death. This will include assisting couples to work together to prepare a will, choose a guardian, and make a financial plan. By focusing on the cost of educating existing children and on the need to plan for their future care, couples are encouraged to reflect on the implications of future childbearing. The interventions will be compared with a standard family planning program with respect to impact on incident pregnancy, contraceptive choice and pattern of use, psychosocial and behavioral variables, and future planning actions. Cost-effectiveness will be determined with methods developed jointly by experts in the fields of HIV therapy in Africa and contraception.

Participants in this study will be randomized to either the user-independent contraception intervention, the future planning intervention, the contraception plus planning intervention, or the standard family planning control. Couples will be followed for 1 to 4 years. Women will have study visits every 3 months; men will have a study visit every year. The primary study outcome will be comparison of time to pregnancy across intervention groups.

ELIGIBILITY:
Inclusion Criteria

* Couples with one or both partners with HIV infection

Exclusion Criteria

* Pregnant or < 1 month post-partum (couples will be invited to return when the infant is > 1 month old)
* Peri- or post-menopausal
* Surgical sterilization or hysterectomy
* Documented infertility

Ages: 16 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5000
Dates: Start 2002-01

PRIMARY OUTCOMES:
pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Susan Allen, MD, MPH, Principal Investigator — Emory University, Rollins School of Public Health
Locations (1):
- Zambia Emory HIV Research Project, Lusaka, Zambia

REFERENCES:
- [Derived] Wall KM, Haddad L, Vwalika B, Htee Khu N, Brill I, Kilembe W, Stephenson R, Chomba E, Vwalika C, Tichacek A, Allen S. Unintended pregnancy among HIV positive couples receiving integrated HIV counseling, testing, and family planning services in Zambia. PLoS One. 2013 Sep 30;8(9):e75353. doi: 10.1371/journal.pone.0075353. eCollection 2013. PMID 24098692
- [Derived] Haddad L, Wall KM, Vwalika B, Khu NH, Brill I, Kilembe W, Stephenson R, Chomba E, Vwalika C, Tichacek A, Allen S. Contraceptive discontinuation and switching among couples receiving integrated HIV and family planning services in Lusaka, Zambia. AIDS. 2013 Oct;27 Suppl 1(0 1):S93-103. doi: 10.1097/QAD.0000000000000039. PMID 24088689
- [Derived] Wall KM, Vwalika B, Haddad L, Khu NH, Vwalika C, Kilembe W, Chomba E, Stephenson R, Kleinbaum D, Nizam A, Brill I, Tichacek A, Allen S. Impact of long-term contraceptive promotion on incident pregnancy: a randomized controlled trial among HIV-positive couples in Lusaka, Zambia. J Acquir Immune Defic Syndr. 2013 May 1;63(1):86-95. doi: 10.1097/QAI.0b013e31827ee19c. PMID 23202814